CLINICAL TRIAL: NCT02179398
Title: Impact of the Lab-score on Antibiotic Prescription Rate in Children Aged 7 Days to 3 Years Old With Fever Without Source.
Brief Title: Impact of the Lab-score on Antibiotic Prescription Rate in Children With Fever Without Source
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Principal Investigator, Laurence Lacroix, Dr, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-162 (MatPed 09-032)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Fever Without Source
Keywords: Fever without source; Antibiotic prescription; Serious bacterial infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lab-score group (Experimental): Patients assessed through the Lab-score determination only: Lab-score ≥3 used as the sole marker for the detection of serious bacterial infection.
  (WBC and band counts blinded to the physician in charge of the patient)
  Interventions: Biological: Allocation to the Lab-score group
- Control group (Active Comparator): Patients assessed through the following classically admitted biomarkers for the detection of serious bacterial infection: WBC count, band count and CRP determination.
  (PCT and thus Lab-score blinded to the physician in charge of the patient).
  Interventions: Biological: Allocation to the control group

INTERVENTIONS:
Biological: Allocation to the Lab-score group
  Arms: Lab-score group
Biological: Allocation to the control group
  Arms: Control group

SUMMARY:
Detecting serious bacterial infections (SBI) in children presenting to the Pediatric Emergency Department (PED) with fever without source (FWS) is a frequent diagnostic challenge. The recently described Lab-score, based on the combined determination of Procalcitonin, C-Reactive Protein (CRP) and urine dipstick results, has been shown an accurate tool for SBI prediction on retrospective cohorts. The investigators aimed to assess the usefulness of the Lab-score in safely decreasing unnecessary antibiotic prescriptions in children with FWS, and to prospectively determine the diagnostic characteristics of the Lab-score compared to other classically used SBI biomarkers (white blood cell (WBC) count, band count and CRP).

ELIGIBILITY:
Inclusion Criteria:

* children aged 7 days to 3 years old
* fever without source ≥ 100.4°F (≥ 38.0°C)

Exclusion Criteria:

* antibiotics received in the previous 48 hours
* underlying congenital or acquired immunodeficiency syndrome
* fever for more than 7 days at presentation

Ages: 7 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence E Lacroix, Principal Investigator — Children's Hospital, Geneva University Hospital
Locations (1):
- Children's Hospital, Geneva University Hospital, Geneva, Geneva 14, Switzerland

REFERENCES:
- [Background] Lacour AG, Zamora SA, Gervaix A. A score identifying serious bacterial infections in children with fever without source. Pediatr Infect Dis J. 2008 Jul;27(7):654-6. doi: 10.1097/INF.0b013e318168d2b4. PMID 18536624
- [Background] Galetto-Lacour A, Zamora SA, Andreola B, Bressan S, Lacroix L, Da Dalt L, Gervaix A. Validation of a laboratory risk index score for the identification of severe bacterial infection in children with fever without source. Arch Dis Child. 2010 Dec;95(12):968-73. doi: 10.1136/adc.2009.176800. Epub 2010 Jun 1. PMID 20515973
- [Background] Bressan S, Gomez B, Mintegi S, Da Dalt L, Blazquez D, Olaciregui I, de la Torre M, Palacios M, Berlese P, Ruano A. Diagnostic performance of the lab-score in predicting severe and invasive bacterial infections in well-appearing young febrile infants. Pediatr Infect Dis J. 2012 Dec;31(12):1239-44. doi: 10.1097/INF.0b013e318266a9aa. PMID 22760529
- [Derived] Lacroix L, Manzano S, Vandertuin L, Hugon F, Galetto-Lacour A, Gervaix A. Impact of the lab-score on antibiotic prescription rate in children with fever without source: a randomized controlled trial. PLoS One. 2014 Dec 11;9(12):e115061. doi: 10.1371/journal.pone.0115061. eCollection 2014. PMID 25503770

RESULTS

PARTICIPANT FLOW:
Groups:
- Lab-score Group: Patients assessed through the Lab-score determination only: Lab-score ≥3 used as the sole marker for the detection of serious bacterial infection.
  (WBC and band counts blinded to the physician in charge of the patient)
  Allocation to the Lab-score group
- Control Group: Patients assessed through the following classically admitted biomarkers for the detection of serious bacterial infection: WBC count, band count and CRP determination.
  (PCT and thus Lab-score blinded to the physician in charge of the patient).
  Allocation to the control group
Period: Overall Study
Arm/Group | Lab-score Group | Control Group
Started | 134 | 144
Completed | 131 | 140
Not Completed | 3 | 4
Not completed — Lack of obligatory data | 3 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lab-score Group | Control Group | Total
Number analyzed (Participants) | 131 | 140 | 271
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 4.8 [1.7 to 10.4] | 3.4 [1.5 to 10.4] | 4.0 [1.6 to 10.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 69 | 135
  Male | 65 | 71 | 136
Fever duration [Number; unit: participants]
  < 12 hours | 47 | 55 | 102
  12-24 hours | 25 | 24 | 49
  > 24 hours | 59 | 61 | 120
Maximum temperature [Mean (Standard Deviation); unit: °C] | 39.3 (0.8) | 39.3 (0.8) | 39.3 (0.78)
Lab-score value [Mean (Standard Deviation); unit: units on a scale] — Lab-score value ranges from 0 to 9. A cutoff point ≥3 was identified as the best Lab-score value for SBI prediction in the original derivation study. A child with a Lab-score < 3 has a low SBI risk, whereas a child with a Lab-score value ≥3 has a high >SBI risk.
  units on a scale | 2.03 (2.62) | 2.04 (2.86) | 2.04 (2.74)
Presence of Serious Bacterial Infection (SBI) [Number; unit: participants] — SBI was defined as isolation of a bacterial pathogen from the blood, the urine, the cerebrospinal fluid, the synovial fluid, the bone, the stools, or by presence of pneumonia (defined as presence of fever, ≥38°C or ≥100.4°F, cough, tachypnea, and a radiographic lung infiltrate).
  participants | 32 | 35 | 67

OUTCOME MEASURES:

1. Primary Outcome: Antibiotic Prescription Rate
Time Frame: at PED (Pediatric Emergency Department) presentation
Population: children 7 days - 36 months old presenting to the PED with fever without source (FWS) ≥38.0°C (≥ 100.4°F) after a thorough history and careful examination
Measure: Number; unit: participants
Groups:
- Lab-score Group: Patients assessed through the Lab-score determination only: Lab-score ≥3 used as the sole marker for the detection of serious bacterial infection.
  (white blood cell (WBC) and band counts blinded to the physician in charge of the patient)
  Allocation to the Lab-score group
- Control Group: Patients assessed through the following classically admitted biomarkers for the detection of serious bacterial infection: white blood cell (WBC) count, band count and C-Reactive Protein (CRP) determination.
  (Procalcitonin (PCT) and thus Lab-score blinded to the physician in charge of the patient).
  Allocation to the control group
Arm/Group | Lab-score Group | Control Group
Number analyzed (Participants) | 131 | 140
participants | 54 | 59
Statistical Analysis 1: Comparison: Lab-score Group vs Control Group; Test type: Superiority or Other; p = 1, Chi-squared

2. Secondary Outcome: Presence of Serious Bacterial Infection
Time Frame: at 72 hours from PED presentation
Measure: Number; unit: participants
Arm/Group | Lab-score Group | Control Group
Number analyzed (Participants) | 131 | 140
participants | 32 | 35
Statistical Analysis 1: Comparison: Lab-score Group vs Control Group; Test type: Superiority or Other; p = 1, Chi-squared

3. Secondary Outcome: Hospitalization Rate
Time Frame: at PED presentation
Measure: Number; unit: participants
Arm/Group | Lab-score Group | Control Group
Number analyzed (Participants) | 131 | 140
participants | 44 | 50
Statistical Analysis 1: Comparison: Lab-score Group vs Control Group; Power calculation suggested 97 patients should be enrolled in each group to give 80% power at the 5% level of significance to detect a 20% difference in antibiotic prescription rate; Test type: Superiority or Other; p = 0.810, Chi-squared

4. Secondary Outcome: Sensitivity of a Lab-score ≥ 3
Time Frame: at 72 hours from PED presentation
Measure: Number (95% Confidence Interval); unit: percentage of patients (sensitivity)
Groups:
- Patients 0-3 Years Old: Patients allocated to the Lab-score group OR to the control group, aged 0 up to 36 months-old.
- Patients < 3 Months Old: Patients allocated to the Lab-score group OR to the control group, aged less than 3 months-old.
Arm/Group | Patients 0-3 Years Old | Patients < 3 Months Old
Number analyzed (Participants) | 271 | 117
percentage of patients (sensitivity) | 85.1 [76.5 to 93.6] | 80.0 [65.7 to 94.3]

5. Secondary Outcome: Specificity of a Lab-score ≥ 3
Time Frame: at 72 hours from PED presentation
Measure: Number (95% Confidence Interval); unit: percentage of patients (specificity)
Arm/Group | Patients 0-3 Years Old | Patients < 3 Months Old
Number analyzed (Participants) | 271 | 117
percentage of patients (specificity) | 87.3 [82.7 to 91.8] | 93.1 [87.8 to 98.4]

6. Secondary Outcome: Sensitivity of Standard Biological Marker for SBI
Description: Sensitivity of standard biological marker for SBI: WBC ≥ 15'000/mm³ and/or bands ≥ 1'500/mm³ and/or CRP ≥ 40 mg/L
Time Frame: at 72 hours from PED presentation
Measure: Number (95% Confidence Interval); unit: percentage of patients (sensitivity)
Arm/Group | Patients 0-3 Years Old | Patients < 3 Months Old
Number analyzed (Participants) | 271 | 117
percentage of patients (sensitivity) | 83.6 [74.7 to 92.5] | 70.0 [53.6 to 86.4]

7. Secondary Outcome: Specificity of Standard Biological Marker for SBI
Description: Specificity of standard biological marker for SBI: WBC ≥ 15'000/mm³ and/or bands ≥ 1'500/mm³ and/or CRP ≥ 40 mg/L
Time Frame: at 72 hours from PED presentation
Measure: Number (95% Confidence Interval); unit: percentage of patients (specificity)
Arm/Group | Patients 0-3 Years Old | Patients < 3 Months Old
Number analyzed (Participants) | 271 | 117
percentage of patients (specificity) | 68.8 [62.4 to 75.2] | 79.3 [70.8 to 87.8]

ADVERSE EVENTS:
Arm/Group | Lab-score Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/140
Other Adverse Events (participants affected / at risk) | 0/131 | 0/140

LIMITATIONS AND CAVEATS:
* heterogeneity in the total number of participating physicians (30)
* recruitment in a tertiary care center (recruitment bias)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No